CLINICAL TRIAL: NCT03923153
Title: Effectiveness of Inspiratory Muscle Training in Patient With Stable Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Irem Hüzmeli, lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MustafaKU 2
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Angina, Stable
Keywords: inspiratory muscle trainig; quality of life; aerobic capacity; depression; fatique
MeSH Terms: conditions — Angina, Stable; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Active Comparator): Inspiratory muscle training group received inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device
  Interventions: Device: Inspiratory muscle training with PowerBreathe (IMT Technologies Ltd., Birmingham,England)
- Sham group (Sham Comparator): Sham group received inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device
  Interventions: Device: Sham group with PowerBreathe (IMT Technologies Ltd., Birmingham, England)

INTERVENTIONS:
Device: Inspiratory muscle training with PowerBreathe (IMT Technologies Ltd., Birmingham,England) — Treatment group II will receive inspiratory muscle endurance training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 30% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 30% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Arms: Inspiratory muscle training group
Device: Sham group with PowerBreathe (IMT Technologies Ltd., Birmingham, England) — Treatment group II will receive inspiratory muscle endurance training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 10% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 30% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Arms: Sham group

SUMMARY:
Stable angina is a cardiac pathology that adversely affects the quality of life of the patient, which develops as a result of narrowing of the coronary vessels developing in atherosclerotic ground and / or impaired oxygen supply-need balance. Studies widely investigated the effects of exercise training in patients with stable angina. No study investigated the effects of inspiratory muscle training in patients with stable angina.Investigators aimed to investigate the effects of inspiratory muscle training on aerobic exercise capacity, quality of life, depression, peripheral and respiratory (MIP, MEP) muscle strength, pulmonary function, dyspnea, fatigue in stable angina patients.

DETAILED DESCRIPTION:
Patients with stable angina will be included. Primary outcome measurement is inspiratory muscle strength, secondary outcomes are functional exercise capacity, peripheral muscle strength, pulmonary functions, maximal exercise capacity, fatigue, quality of life, depression.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication for pulmonary physiotherapy
* Anjina patients who are clinically stable
* have no other disease that may affect respiratory function
* Individuals who have the good cooperation

Exclusion Criteria:

* Patients under the age of 18
* Pregnancy
* Active infection
* Patients with known malignancies
* patients without consent
* known arrhythmia, dilated or hypertrophic cardiomyopathy, heart failure (EF <40%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change of the Inspiratory and expiratory muscle strength (MIP, MEP) from baseline to 8 week | Baseline, after 8 week
  Mouth pressure device( MicroRPM, Micro Medical England)

SECONDARY OUTCOMES:
Change from Baseline Functional exercise capacity at 8 week | Baseline, after 8 week
  6 minute walking test
Change from Pulmonary functions at 8 week | Baseline, after 8 week
  Spirometry
Fatigue | Baseline, after 8 week
  Change from baseline Fatigue Severity Scale (FSS) (Turkish version of scale) at 8 weeek.
  Patient choose a number from 1 to 7 that indicates how much the patient agrees with each statement, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue
Depression | Baseline,after 8 week
  Change from baseline Montgomery Asberg Depression Rating Scale (MADRS) (Turkish version of scale) at 8 week.
  This assessment tool contains 10 items with a score from 0 to 6, thus the maximum score is 60. A higher score indicates a more severe depression.

OTHER OUTCOMES:
Quality life | Baseline, after 8 week
  Change of baseline quality of life at 8 week .Short Form (SF-36) Health Survey (Turkish version of scale) The SF-36 is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning (10 items) social functioning (2 items) role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items). For each dimension item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).

CONTACTS AND LOCATIONS:
Overall Officials: Aysel yıldız, assoc prof, Study Director — Marmara University Faculty of Health Sciences; Irem Hüzmeli, Msc, Study Chair — Mustafa Kemal University; Oğuz Akkuş, assist prof, Principal Investigator — Mustafa Kemal University; Fatih Yalçın, Prof., Study Chair — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kellens I, Cannizzaro F, Gouilly P, Crielaard JM. [Inspiratory muscles strength training in recreational athletes]. Rev Mal Respir. 2011 May;28(5):602-8. doi: 10.1016/j.rmr.2011.01.008. Epub 2011 Apr 19. French. PMID 21645830
- [Background] Long L, Anderson L, Dewhirst AM, He J, Bridges C, Gandhi M, Taylor RS. Exercise-based cardiac rehabilitation for adults with stable angina. Cochrane Database Syst Rev. 2018 Feb 2;2(2):CD012786. doi: 10.1002/14651858.CD012786.pub2. PMID 29394453
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831